CLINICAL TRIAL: NCT00444275
Title: A Randomized, Open, Parallel-group Study to Evaluate the Efficacy of Three Different Patient Management Strategies During a 12 Weeks Maintenance Phase Following an Initial 4-weeks Acute Treatment Phase in Subjects With Symptoms Thought to be GERD Related
Brief Title: Nexium (Esomeprazole) in Symptom Adapted Therapy in GERD Patients
Acronym: MAESTRO
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D9612L00111; EudraCT No: 2006-002867-19
Record Dates: First submitted 2007-03-05; First posted 2007-03-07 (Estimated); Results first posted 2012-12-11 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-11

CONDITIONS: GERD
Keywords: Gastroesophageal Reflux Disease; Acid Reflux
MeSH Terms: conditions — Gastroesophageal Reflux | interventions — Esomeprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Esomeprazole 20 mg Once Daily (initial phase) (Experimental)
  Interventions: Drug: esomeprazole (Nexium®)
- Esomeprazole 40 mg Once Daily (initial phase) (Experimental)
  Interventions: Drug: esomeprazole (Nexium®)
- Esomeprazole 20 mg Once Daily (Maintenance Phase) (Experimental)
  Interventions: Drug: esomeprazole (Nexium®)
- Esomeprazole 20 mg on Demand (Maintenance Phase) (Experimental)
  Interventions: Drug: esomeprazole (Nexium®)
- Antacid Treatment (Maintenance Phase) (Experimental)
  Interventions: Drug: Xolaam®

INTERVENTIONS:
Drug: esomeprazole (Nexium®) — This randomized study was conducted on parallel groups and included two phases:
  * One initial phase during when the patients received once daily, either esomeprazole 20 mg or esomeprazole 40 mg, depending on the investigator's decision
  * One maintenance treatment phase, patients were randomized to one of the following three groups, either esomeprazole 20 mg once daily, or esomeprazole 20 mg on demand or antacid treatment as needed
  Arms: Esomeprazole 20 mg Once Daily (Maintenance Phase); Esomeprazole 20 mg Once Daily (initial phase); Esomeprazole 20 mg on Demand (Maintenance Phase); Esomeprazole 40 mg Once Daily (initial phase)
Drug: Xolaam® — This randomized study was conducted on parallel groups and included two phases:
  * One initial phase during when the patients received once daily, either esomeprazole 20 mg or esomeprazole 40 mg, depending on the investigator's decision
  * One maintenance treatment phase, patients were randomized to one of the following three groups, either esomeprazole 20 mg once daily, or esomeprazole 20 mg on demand or antacid treatment as needed
  Arms: Antacid Treatment (Maintenance Phase)

SUMMARY:
To compare the efficacy of three different long-term treatment strategies of reflux disease in primary care setting.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who seek medical advice in primary care for symptoms thought to be GERD related (GERD is a condition which develops when the reflux of stomach content causes troublesome symptoms and / or complications).

Exclusion Criteria:

* Subjects with any clinical GERD treatment (PPI, H2-receptor antagonists) within the last 3 months prior to Visit 1.
* A history of severe esophagitis or known other complications, with alarm symptoms

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3029 (Actual)
Dates: Start 2007-03; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca France Medical Director, MD, Study Director — AstraZeneca
Locations (1):
- Research Site, Rouen, France

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited by general practitioner between March 1, 2007 and July 21, 2008
Pre-assignment Details: The study included 2 phases (maximum treatment duration = 16 weeks):
  * one initial treatment phase of 4 weeks
  * one randomized maintenance treatment phase of 12 weeks only for patients whose initial treatment is considered to be successful at the end of the initial phase.
  Only maintenance phase data were reported in the Baseline module measures.
Groups:
- Antacid Treatment (Maintenance Phase): antacid treatment as needed (maintenance phase) (Xolaam® maximum six tablets per day)
Period: Initial Treatment Phase
Arm/Group | Esomeprazole 20 mg Once Daily (Initial Phase) | Esomeprazole 40 mg Once Daily (Initial Phase) | Esomeprazole 20 mg Once Daily (Maintenance Phase) | Esomeprazole 20 mg on Demand (Maintenance Phase) | Antacid Treatment (Maintenance Phase)
Started | 2156 | 873 | 0 | 0 | 0
Completed | 1908 | 777 | 0 | 0 | 0
Not Completed | 248 | 96 | 0 | 0 | 0
Period: Maintenance Treatment Phase
Arm/Group | Esomeprazole 20 mg Once Daily (Initial Phase) | Esomeprazole 40 mg Once Daily (Initial Phase) | Esomeprazole 20 mg Once Daily (Maintenance Phase) | Esomeprazole 20 mg on Demand (Maintenance Phase) | Antacid Treatment (Maintenance Phase)
Started | 0 | 0 | 908 | 897 | 880
Completed | 0 | 0 | 747 | 764 | 701
Not Completed | 0 | 0 | 161 | 133 | 179
Not completed — Didn'r receive the treatment | 0 | 0 | 22 | 17 | 29
Not completed — Lost to Follow-up | 0 | 0 | 8 | 14 | 10
Not completed — Adverse Event | 0 | 0 | 3 | 2 | 13
Not completed — Protocol specific criteria's development | 0 | 0 | 1 | 0 | 6
Not completed — Patient's wish | 0 | 0 | 19 | 9 | 20
Not completed — Protocol Violation | 0 | 0 | 103 | 88 | 87
Not completed — Ineffectiveness | 0 | 0 | 5 | 3 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Esomeprazole 20 mg Once Daily (Maintenance Phase) | Esomeprazole 20 mg on Demand (Maintenance Phase) | Antacid Treatment (Maintenance Phase) | Total
Number analyzed (Participants) | 871 | 857 | 830 | 2558
Age Continuous [Mean (Standard Deviation); unit: years] | 41.5 (9.83) | 41.79 (9.97) | 41.6 (10) | 41.64 (9.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 449 | 415 | 411 | 1275
  Male | 422 | 442 | 419 | 1283

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Three Strategies of Long-term Treatment
Description: Percentage of failure of maintenance treatment between V2 (4 weeks) and V3 (16 weeks) evaluated by the patient, defined based on responses to 2 questions (if at least 1 negative response was given, the patient was considered to be in failure) : Did the treatment produce sufficient control of reflux symptoms? Do you wish to continue the treatment?
Time Frame: 16 weeks
Measure: Number; unit: Percentage of participants with failure
Arm/Group | Esomeprazole 20 mg Once Daily (Maintenance Phase) | Esomeprazole 20 mg on Demand (Maintenance Phase) | Antacid Treatment (Maintenance Phase)
Number analyzed (Participants) | 871 | 857 | 830
Percentage of participants with failure | 10.6 | 7.8 | 43

2. Secondary Outcome: Difference in Symptom Severity Evaluation Performed by the Investigators, When Symptom Severity is Assessed With and Without Reflux Disease Questionnaire (RDQ).
Description: Total percentage of subjects for whom evaluation of symptom severity using the Reflux Disease Questionnaire (RDQ) is different, either positively or negatively, as compared to clinical judgment made by Investigator.
  The RDQ Includes 12 Items: 6 Concern the Frequency of Symptoms Ranging From "Never" for the Lowest Frequency to "Every Day" for the Highest, 6 Others Assess the Severity of Symptoms From "Not at All" to "Strong". The Total Score of the RDQ, Ranging From 0 to 40, is Obtained by Adding the Scores of Each Item.
Time Frame: 4 weeks
Measure: Number; unit: Percentage of participants
Arm/Group | Esomeprazole 20 mg Once Daily (Initial Phase) | Esomeprazole 40 mg Once Daily (Initial Phase) | Esomeprazole 20 mg Once Daily (Maintenance Phase) | Esomeprazole 20 mg on Demand (Maintenance Phase) | Antacid Treatment (Maintenance Phase)
Number analyzed (Participants) | 1909 | 778 | 0 | 0 | 0
Percentage of participants | 3.7 | 2.3 |  |  |

3. Secondary Outcome: Impact of Treatment With Low Dose Aspirin (Acetyl Salicylic Acid) Used Concomitantly During the Initial Phase and the Maintenance Phase
Description: No possibility to describe as only 2 patients took ASA
Time Frame: 4 weeks
Population: Outcome measure not possible to describe as only 2 patients took Aspirin.
Arm/Group | Esomeprazole 20 mg Once Daily (Initial Phase) | Esomeprazole 40 mg Once Daily (Initial Phase) | Esomeprazole 20 mg Once Daily (Maintenance Phase) | Esomeprazole 20 mg on Demand (Maintenance Phase) | Antacid Treatment (Maintenance Phase)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Differences Among Strategies of Maintenance Treatment for Satisfaction of the Patient, Using the GIS (Gord Impact Scale) Scale.(Change in Values of Score Derived From the GIS Questionnaire From V2 to V3 = Start to End of the Maintenance Phase)
Description: Change in values of upper digestive symptoms (GORD Impact Scale) from week 4 to week 16. Scale of 1 to 4 : 1 = every day, 2 = often, 3 = sometime, 4 = never)
Time Frame: 4 to 16 weeks
Population: 871 (-66 missing data, 801 (-56 missing data), 833 (-75 missing data)
Measure: Mean (Standard Deviation); unit: Scores on scale
Arm/Group | Esomeprazole 20 mg Once Daily (Initial Phase) | Esomeprazole 40 mg Once Daily (Initial Phase) | Esomeprazole 20 mg Once Daily (Maintenance Phase) | Esomeprazole 20 mg on Demand (Maintenance Phase) | Antacid Treatment (Maintenance Phase)
Number analyzed (Participants) | 0 | 0 | 871 | 801 | 833
Scores on scale |  |  | 0.12 (0.79) | 0.04 (0.73) | -0.22 (0.8)

5. Secondary Outcome: Impact of Anxiety and Depression During the Initial Visit Measured by the HADS ( Hospital Anxiety and Depression Scale) Questionnaire on Response to Initial Treatment and to Maintenance Treatment
Description: Failure of treatment (as defined as in primary outcome measure) according to confirmed anxiety and depression during maintenance treatment evaluated by the patient via the score of HADS questionnaire. HADS scale ranges= 0 to 21 (the higher score, the worse : ≤7 : no anxiety-depression/ [8-10] : possible anxiety-depression/ >10 : anxiety-depression)
Time Frame: 16 weeks
Measure: Number; unit: Percent of participants with failure
Arm/Group | Esomeprazole 20 mg Once Daily (Initial Phase) | Esomeprazole 40 mg Once Daily (Initial Phase) | Esomeprazole 20 mg Once Daily (Maintenance Phase) | Esomeprazole 20 mg on Demand (Maintenance Phase) | Antacid Treatment (Maintenance Phase)
Number analyzed (Participants) | 0 | 0 | 871 | 857 | 830
Percent of participants with failure |  |  | 9.8 | 9.3 | 43.7

6. Secondary Outcome: Number of Participants and Type of Serious Adverse Events and Adverse Events Leading to a Premature Discontinuation of the Study
Description: Number of participants with serious adverse events and adverse events leading to study treatment discontinuation. AE and SAE as defined in ICH-GCP.
Time Frame: 12 weeks - maintenance treatment phase
Measure: Number; unit: Participants
Arm/Group | Esomeprazole 20 mg Once Daily (Initial Phase) | Esomeprazole 40 mg Once Daily (Initial Phase) | Esomeprazole 20 mg Once Daily (Maintenance Phase) | Esomeprazole 20 mg on Demand (Maintenance Phase) | Antacid Treatment (Maintenance Phase)
Number analyzed (Participants) | 0 | 0 | 886 | 880 | 851
Participants |  |  | 5 | 4 | 15

7. Secondary Outcome: Score Abacuses Based on the Reflux Disease Questionnaire (RDQ) Questionnaire
Description: May be used to evaluate the severity of symptoms during the initial visit. Not done
Time Frame: Day 0
Population: The results of exploratory analyses are not available.
Arm/Group | Esomeprazole 20 mg Once Daily (Initial Phase) | Esomeprazole 40 mg Once Daily (Initial Phase) | Esomeprazole 20 mg Once Daily (Maintenance Phase) | Esomeprazole 20 mg on Demand (Maintenance Phase) | Antacid Treatment (Maintenance Phase)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Score Abacuses Based on the Reflux Disease Questionnaire (RDQ) Questionnaire
Description: May be used to offer patients a strategy of treatment during the initial phase and in the long term.
  Not done
Time Frame: Day 0
Population: The results of exploratory analyses are not available.
Arm/Group | Esomeprazole 20 mg Once Daily (Initial Phase) | Esomeprazole 40 mg Once Daily (Initial Phase) | Esomeprazole 20 mg Once Daily (Maintenance Phase) | Esomeprazole 20 mg on Demand (Maintenance Phase) | Antacid Treatment (Maintenance Phase)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Score Abacuses Based on the Reflux Disease Questionnaire (RDQ)
Description: May be used to define the success of treatment. Not done
Time Frame: Week 4
Population: The results of exploratory analyses are not available.
Arm/Group | Esomeprazole 20 mg Once Daily (Initial Phase) | Esomeprazole 40 mg Once Daily (Initial Phase) | Esomeprazole 20 mg Once Daily (Maintenance Phase) | Esomeprazole 20 mg on Demand (Maintenance Phase) | Antacid Treatment (Maintenance Phase)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Esomeprazole 20 mg Once Daily (Initial Phase) | Esomeprazole 40 mg Once Daily (Initial Phase) | Esomeprazole 20 mg Once Daily (Maintenance Phase) | Esomeprazole 20 mg on Demand (Maintenance Phase) | Antacid Treatment (Maintenance Phase)
Serious Adverse Events (participants affected / at risk) | 8/2156 | 2/873 | 2/886 | 3/880 | 4/851
Other Adverse Events (participants affected / at risk) | 32/2156 | 16/873 | 5/886 | 2/880 | 13/851
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Esomeprazole 20 mg Once Daily (Initial Phase) (N=2156) | Esomeprazole 40 mg Once Daily (Initial Phase) (N=873) | Esomeprazole 20 mg Once Daily (Maintenance Phase) (N=886) | Esomeprazole 20 mg on Demand (Maintenance Phase) (N=880) | Antacid Treatment (Maintenance Phase) (N=851)
ACUTE BALTHAZAR E PANCREATITIS (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
GASTRIC ULCER (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
ANXIO-DEPRESSI VE STATE (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
AGGRAVATION OF INTERVERTEBRAL DISC HERNIATION (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0
RENAL COLIC (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 1
EROSIVE ANTRITIS (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
BRONCHIAL CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
SPONDYLOLISTHE SIS AGGRAVATION BY L5 SPONDYLOLYSIS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
DEPRESSION (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0
PNEUMOPATHY (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
ADENOCARCINOM A OF GASTRIC ANTRUM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
DIGESTIVE VIROSIS (Infections and infestations) | 0 | 0 | 0 | 1 | 0
DEPRESSIVE DISEASE (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
CARCINOMA OF OESOPHAGUS (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
PREEXISTING LUNG CARCINOMA AGGRAVATION (General disorders) | 1 | 0 | 0 | 0 | 0
ADENOMATOUS POLYP (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
METRORRHAGIA (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Esomeprazole 20 mg Once Daily (Initial Phase) (N=2156) | Esomeprazole 40 mg Once Daily (Initial Phase) (N=873) | Esomeprazole 20 mg Once Daily (Maintenance Phase) (N=886) | Esomeprazole 20 mg on Demand (Maintenance Phase) (N=880) | Antacid Treatment (Maintenance Phase) (N=851)
Dyspepsia (Vascular disorders) | 2 | 2 | 1 | 1 | 3
Diarrhea (Gastrointestinal disorders) | 3 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 5 | 2 | 1 | 0 | 0
Epigastric discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 1 | 0 | 0 | 0
Chest pain (General disorders) | 0 | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 4 | 1 | 0 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 3 | 1 | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 2 | 0 | 0 | 0
Pharyngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Somnolence (General disorders) | 1 | 0 | 0 | 0 | 0
Weight decreased (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Nervousness (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Planned number of patients not reached: statistical analysis plan revised,comparisons between treatment arms performed globally (No stratified analysis).

Safety pop=3032-3 incorrect enrolments (withdrawals at V2) with no information on ttmt received

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No